CLINICAL TRIAL: NCT01215071
Title: Prospektiv Randomisierte Studie Zum Vergleich Einer Ausgedehnten Mit Einer eingeschränkten Pelvinen Lymphadenektomie Bei Der Operativen Therapie Des Harnblasenkarzinoms
Brief Title: Eingeschränkte vs Ausgedehnte Lymphadenektomie LEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association of Urologic Oncology (AUO) (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB 25/02
Record Dates: First submitted 2010-09-29; First posted 2010-10-06 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Bladder Cancer
Keywords: Lymphadenectomy; Extension; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- limited lymphadenectomy (Experimental): Fields 5, 7, 9, 11, 13, 14 are removed
  Interventions: Procedure: limited lymphadenectomy
- extended lymphadenectomy (Experimental): Fields 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 are removed
  Interventions: Procedure: extended lymphadenectomy

INTERVENTIONS:
Procedure: limited lymphadenectomy — Field 5 (Group external iliac rigt) Field 7 (Group external iliac left) Field 9 (obturatorical Group right) Field 11 (obturatorical Group left) Field 13 (Group internal iliac right) Field 14 (Group internal iliac left)
  Other Names: eingeschränkte Lymphadenektomie; eingeschränkte LA
  Arms: limited lymphadenectomy
Procedure: extended lymphadenectomy — Field 1 (paracaval right) Field 2 (interaortocaval) Field 3 (paraaortal left) Field 4 (Group iliac artery right) Field 5 (Group external iliac rigt) Field 6 (Group iliac artery left) Field 7 (Group external iliac left) Field 8 (presacral) Field 9 (obturatorical Group right) Field 10 (deep obturatorical Group right) Field 11 (obturatorical Group left) Field 12 (deep obturatorical Group left) Field 13 (Group internal iliac right) Field 14 (Group internal iliac left)
  Other Names: ausgedehnte Lymphadenektomie; ausgedehnte LA
  Arms: extended lymphadenectomy

SUMMARY:
This trial evaluates the therapeutic benefit of extended versus limited lymphadenectomy at the time of radical cystectomy in patients with bladder cancer.

DETAILED DESCRIPTION:
The extent of pelvic lymphadenectomy in the surgical treatment of muscle-invasive, clinically locally bladder cancer is not yet standardized. There are no data from randomized, prospective studies on the prognostic role of regional lymphadenectomy.

Results of retrospective studies suggest, that the prognosis of patients with muscle-invasive bladder cancer can be improved by extending the limits of pelvic lymphadenectomy. Furthermore it could be demonstrated in a prospective study that the pattern of metastasis of bladder cancer has a high variability. About two-thirds of lymph node metastases are found outside the normally cleared areas of lymphadenectomy. In this study patients will be randomized into arms with limited versus extended lymphadenectomy.

The limited lymphadenectomy includes the removal of the obturatoric, external and internal iliac lymph nodes, the extended one includes the removal of all lymph nodes between pelvic floor and the inferior mesenteric artery. The primary objective of the study is to detemine the influence of limited versus extended lyphadenectomy at the time of radical cystectomy on recurrence-free survival. Secondary study objectives include the influence on cancer-specific survival, overall survival, complication rates, histopathologic N-stage, the localization of recurrence and influence of adjuvant chemotherapy . Adjuvant chemotherapy is optional and is recommended in patients with locally advanced disease (pT3/4) or regional lymph node metastasis (pN+).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, invasive urothelial bladder cancer, locally completely resectable (T1G3 - T4a, Nx)
* Age >= 18 years
* Written consent of the patient
* Patient compliance and geographic proximity to allow adequate follow-up

Exclusion Criteria:

* Histologically or by imaging diagnostics proven organ metastases
* Radiographic evidence of enlarged lymph nodes (> 1 cm) above the aortic bifurcation in conjunction with pelvic lymph node metastases
* Radiographic or other evidence of T4b-tumor (infiltration of the pelvic wall or other organ systems)
* Prior neoadjuvant chemotherapy of bladder cancer
* Prior previous pelvic lymphadenectomy
* Prior radiotherapy to the pelvis
* internal medical or anesthetic risk factors that require a short operation time
* Palliative cystectomy (f.e. bulky-disease, infiltration of adjacent structures)
* Evidence of another tumor restricting life expectancy of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2006-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Recurrence free Survival (RFS) | 5 years
  Definition Recurrence-free survival: Time from radical cystectomy to tumor reccurence or death from any cause up to 5 years

SECONDARY OUTCOMES:
Cancer specific survival (CSS) | 5 years
  Definition Cancer-specific suvival: Time from radical cystectomy to death from bladder cancer up to 5 years
Overall survival (OS) | 5 years
  Definition Overall survival: Time from radical cystectomy to death from any cause up to 5 years
Determination of type and location of tumour progression(local recurrences and distant metastases) | 5 years
Effect on histopathological stage (Will Rogers phenomenon) | 5 years
  Definition Effect on histopathologic stage: Influence of extended lymphadenectomy on detection of lymph node metastasis
Influence of adjuvant chemotherapy (by subgroup analysis) | 5 years
Documentation of complications | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen E. Gschwend, Prof. Dr., Principal Investigator — AUO - Association of Urologic Oncology
Locations (16):
- Germany (16):
  - University of Cologne, Cologne
  - Hospital Holweide, Cologne
  - Urological hospital, Städt. Kliniken Dortmund, Dortmund
  - Paracelsus Hospital, Düsseldorf
  - Heinrich Heine University, Düsseldorf
  - University of Essen, Essen
  - Department of urology, städt. Klinikum Fulda, Fulda
  - Saarland University, Homburg/Saar
  - Städt. Klinikum, Karlsruhe
  - Urological Hospital Kassel, Kassel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Otto von Guericke University, Magdeburg
  - Klinikum r. d. Isar der TUM, München
  - Eberhard Karls University, Tübingen
  - Urological hospital, University Hospital Ulm, Ulm
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Gschwend JE, Heck MM, Lehmann J, Rubben H, Albers P, Wolff JM, Frohneberg D, de Geeter P, Heidenreich A, Kalble T, Stockle M, Schnoller T, Stenzl A, Muller M, Truss M, Roth S, Liehr UB, Leissner J, Bregenzer T, Retz M. Extended Versus Limited Lymph Node Dissection in Bladder Cancer Patients Undergoing Radical Cystectomy: Survival Results from a Prospective, Randomized Trial. Eur Urol. 2019 Apr;75(4):604-611. doi: 10.1016/j.eururo.2018.09.047. Epub 2018 Oct 15. PMID 30337060
- [Derived] Froehner M, Novotny V, Heberling U, Rutsch L, Litz RJ, Hubler M, Koch R, Baretton GB, Wirth MP. Relationship of the number of removed lymph nodes to bladder cancer and competing mortality after radical cystectomy. Eur Urol. 2014 Dec;66(6):987-90. doi: 10.1016/j.eururo.2014.07.046. Epub 2014 Aug 19. PMID 25150172
- See also: The AUO Homepage where this study is presented — http://www.auo-online.de